CLINICAL TRIAL: NCT03504982
Title: Study to Clinically Evaluate the QT/QTc Interval Prolongation Potential of Vericiguat in Patients With Stable Coronary Artery Disease in a 2-arm, Placebo-controlled, Randomized, Double-blind, Double-dummy Design Including a Vericiguat Multiple-dose Part With Fixed up Titration Periods and Moxifloxacin as Positive Control (for Assay Sensitivity Testing, Nested Into the Placebo Treatment)
Brief Title: Study to Evaluate the QT / QTc Interval Prolongation Potential of Vericiguat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18979; 2017-003094-33 (EudraCT Number)
Record Dates: First submitted 2018-04-13; First posted 2018-04-20 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease
Keywords: Vericiguat; Stable CAD; QT/QTc
MeSH Terms: conditions — Coronary Artery Disease | interventions — vericiguat; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment 1 (Experimental): Treatment sequences: A*-B-C-D
  Interventions: Drug: Vericiguat (BAY1021189); Drug: Moxifloxacin; Drug: Placebo
- Treatment 2 (Experimental): Treatment sequences: D-A-B-C*
  Interventions: Drug: Vericiguat (BAY1021189); Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) — A : 2.5 mg vericiguat A*: 2.5 mg vericiguat B : 5 mg vericiguat C : 10 mg vericiguat C*: 10 mg vericiguat
Drug: Moxifloxacin — D: 400 mg moxifloxacin
Drug: Placebo — A : vericiguat placebo 10 mg A*: vericiguat placebo 10 mg + moxifloxacin placebo B : vericiguat placebo 10 mg C : vericiguat placebo 2.5 mg C*: vericiguat placebo 2.5 mg + moxifloxacin placebo D : vericiguat placebo 2.5 mg + vericiguat placebo 10 mg

SUMMARY:
The primary objective of this study was to investigate whether there is a clinically meaningful effect on QTc change from baseline relative to placebo after administration of 10 mg at steady state in patients with stable CAD (coronary artery disease).

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable CAD (coronary artery disease) defined by:

  * clinically stable for at least 3 months
  * coronary artery stenosis in any of the 3 main coronary vessels
  * or history of myocardial infarction
* Sinus rhythm at screening
* Interpretable echocardiographic images
* Age: 30 to 80 years
* Body mass index (BMI): above/equal 18.0 and below/equal 36.0 kg/m²

Exclusion Criteria:

* Ejection fraction (EF) below 30% at screening
* Progressive angina with symptoms of worsening of angina within the <3 month
* History of recent myocardial infarction or unstable Angina
* Documented current relevant coronary stenosis ≥90% in any of the main 3 coronary vessels without bypass graft
* Symptomatic carotid stenosis, or transient ischemic attack or stroke within 3 months or patients with stroke at more than 3 months
* Insulin dependent diabetes mellitus
* Clinically significant and persisting cardiac ischemia
* Atrial fibrillation, pacemaker, defibrillator, second and third degree atrial-ventricular (AV) block
* Known clinically relevant ventricular arrhythmias
* Clinically relevant heart failure with reduced left ventricular ejection fraction
* Significant valvular heart disease with moderate or severe aortic stenosis or any other significant stenosis; any other moderate or severe valvular failures
* Valve replacement
* Hypertrophic obstructive cardiomyopathy (HOCM)
* Previous or imminent cardiac transplantation
* Known long QT syndrome or prolongation of the QT interval with ongoing proarrhythmic conditions
* Co-medication with drugs known to have QT prolonging effect
* Intolerance of fluoroquinolones, including moxifloxacin
* History of serious adverse effects e.g. tendinitis and tendon rupture, arthralgia and effects on the peripheral and central nervous system while taking fluoroquinolones including moxifloxacin
* History of tendon diseases or tendon injury caused by quinolones
* Treatment with fluoroquinolones, including moxifloxacin during the last 2 weeks
* Treatment with organic nitrates during the last 3 months
* Treatment with riociguat during the last 3 months
* Treatment with phosphodiesterase (PDE)-5 inhibitors during the last 14 days
* Systolic blood pressure below 110 or above 160 mmHg at screening visit
* Diastolic blood pressure below 50 or above 100 mmHg at screening visit
* Heart rate below 50 or above 100 beats/min (taken from ECG measurement) at first screening visit
* Estimated glomerular filtration rate (eGFR) below 30 mL/min/1.73m*2

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Time-matched placebo-corrected change from baseline of the QT interval corrected according to Fridericia (QTcF) after 10 mg vericiguat at steady state. | Baseline, day 56 (steady state 10 mg) of vericiguat treatment

SECONDARY OUTCOMES:
Time-matched placebo-corrected change from baseline of QTcF after 1st dose of 2.5 mg vericiguat | Baseline and day 1 of vericiguat treatment
Time-matched placebo-corrected change from baseline of QTcF after 1st dose of 5 mg vericiguat | Baseline and day 15 (+/- 3 days) of vericiguat treatment
Time-matched placebo-corrected change from baseline of QTcF after 1st dose of 10 mg vericiguat | Baseline and day 29 (+/- 3 days) of vericiguat treatment
Time-matched placebo-corrected change from baseline of QTcF after 2.5 mg vericiguat at steady state | Baseline and day 14 (+/- 3 days) of vericiguat treatment (steady state 2.5 mg)
Time-matched placebo-corrected change from baseline of QTcF after 5 mg vericiguat at steady state | Baseline and day 28 (+/- 3 days) of vericiguat treatment (steady state 5 mg)
Time-matched placebo-corrected change from baseline of QTcF after single dose of moxifloxacin | Baseline and day 8 of the moxifloxacin treatment period
Maximum concentration of vericiguat in plasma after first dose (Cmax) | On profile day 1; Timeframe: 0 - 5 hours after dosing
Time to maximum concentration of vericiguat in plasma after first dose (tmax) | On profile day 1; Timeframe: 0 - 5 hours after dosing
Maximum concentration of vericiguat in plasma after multiple doses (Cmax, md) | On profile days: 8, 14, 15, 28, 29, 42, 43, 50 and 56; Timeframe: 0 - 5 hours after dosing
Time to maximum concentration of vericiguat in plasma after multiple doses (tmax, md) | On profile days: 1, 8, 14, 15, 28, 29, 42, 43, 50 and 56; Timeframe: 0 - 5 hours after dosing
Maximum concentration of moxifloxacin in plasma after single dose (Cmax) | On moxifloxacin profile days (day 8 and 50); Timeframe: 0 - 5 hours after dosing
Time to maximum concentration of moxifloxacin in plasma after single dose (tmax) | On moxifloxacin profile days (day 8 and 50); Timeframe: 0 - 5 hours after dosing
Number of subjects with treatment-emergent adverse events (TEAEs) | 12 months

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (6):
  - Universitätsherzzentrum Freiburg - Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Medizinische Einrichtungen der Universität Bonn, Bonn, North Rhine-Westphalia
  - SocraTec R&D Clinical Ward, Erfurt, Thuringia
  - Charité Campus Virchow-Klinikum (CVK), Berlin
  - PAREXEL GmbH, Berlin
- IMSP Republican Clinical Hospital, Chisinau, Moldova
- Center for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Ruehs H, Solms A, Frei M, Becker C, Trujillo ME, Garmann D, Meyer M. Assessing QTc Effects of Vericiguat Using Two Different Concentration-QTc Modeling Approaches. Clin Pharmacokinet. 2023 Nov;62(11):1639-1648. doi: 10.1007/s40262-023-01282-y. Epub 2023 Sep 6. PMID 37672197
- [Derived] Bottcher M, Dungen HD, Corcea V, Donath F, Fuhr R, Gal P, Mikus G, Trenk D, Coenen M, Pires PV, Maschke C, Aliprantis AO, Besche N, Becker C. Vericiguat: A Randomized, Phase Ib, Placebo-Controlled, Double-Blind, QTc Interval Study in Patients with Chronic Coronary Syndromes. Am J Cardiovasc Drugs. 2023 Mar;23(2):145-155. doi: 10.1007/s40256-022-00557-2. Epub 2023 Jan 12. PMID 36633816